CLINICAL TRIAL: NCT04785976
Title: Long-term Prognosis of Emergency Aneurysmal Subarachnoid Hemorrhage: an MDT- Based Multicenter Cohort Study
Brief Title: Long-term Prognosis of Emergency Aneurysmal Subarachnoid Hemorrhage
Acronym: LongTEAM
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Peking University International Hospital (Other)
Responsible Party: Principal Investigator, yuanli Zhao, Director of Department of Cerebrovascular Neurosurgery, Beijing Tiantan Hospital
Other Study IDs: KY 2020-11-26
Record Dates: First submitted 2021-02-01; First posted 2021-03-08 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical clipping
  Interventions: Procedure: Surgical clipping and endovascular coiling
- Endovascular coiling
  Interventions: Procedure: Surgical clipping and endovascular coiling

INTERVENTIONS:
Procedure: Surgical clipping and endovascular coiling — Surgical clipping: Apply aneurysm clip to clip the ruptured aneurysm. Endovascular coiling：Also called endovascular embolization, to block blood flow into an aneurysm.Preventing blood flow into an aneurysm helps to keep it from rupturing.

SUMMARY:
Rupture of intracranial aneurysms can lead to extensive subarachnoid hemorrhage (SAH), a potentially fatal neurological emergency with mortality rates ranging from 8 to 67%. At present, surgical clipping (SC) and endovascular coiling (EC) are two main treatments for aneurysmal subarachnoid hemorrhage (aSAH), in recent years, the improvements in surgical equipment and techniques have already greatly improved the postoperative safety of patients. However, considering individual differences between patients, some still at risk due to possible complications during hospitalization or after discharge from the hospital, it will no doubt generate a large healthcare burden.

This prospective, observational clinical trial (LongTEAM) is to improve the diagnosis and treatment effect and efficiency in this field, reducing mortality, medical costs, and medical burden, while opening up new avenues for interdisciplinary clinical practice and scientific research exploration.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the emergency department of the investigator with aneurysmal subarachnoid hemorrhage are included in their prospective registry.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to the emergency department of the investigator with aneurysmal subarachnoid hemorrhage are included in their prospective registry
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2012-04-01 (Actual); Primary Completion 2032-03-01 (Estimated); Study Completion 2032-04-01 (Estimated)

PRIMARY OUTCOMES:
Unfavorable neurological outcome (mRS>2) | 10 days after the procedure
  Number of patients experiencing a unfavorable neurological outcome at discharge, defined as a modified Rankin Scale (mRS) score of >2.
Unfavorable neurological outcome (mRS>2) | 3 months
  Number of patients experiencing a unfavorable neurological outcome at 3 months post-treatment, defined as a modified Rankin Scale (mRS) score of >2.
Unfavorable neurological outcome (mRS>2) | 6 months
  Number of patients experiencing a unfavorable neurological outcome at 6 months post-treatment, defined as a modified Rankin Scale (mRS) score of >2.
Unfavorable neurological outcome (mRS>2) | 12 months
  Number of patients experiencing a unfavorable neurological outcome at 12 months post-treatment, defined as a modified Rankin Scale (mRS) score of >2.
Unfavorable neurological outcome (mRS>2) | 24 months
  Number of patients experiencing a unfavorable neurological outcome at 24 months post-treatment, defined as a modified Rankin Scale (mRS) score of >2.

SECONDARY OUTCOMES:
Cognitive deficits | 10 days after the procedure
  Number of patients experiencing a unfavorable neurological outcome at discharge,defined as changes in thinking, emotion, will and behavior.
Cognitive deficits | 3 months
  Number of patients experiencing a unfavorable neurological outcome at 3 months, defined as changes in thinking, emotion, will and behavior.
Cognitive deficits | 6 months
  Number of patients experiencing a unfavorable neurological outcome at 6 months, defined as changes in thinking, emotion, will and behavior.
Cognitive deficits | 12 months
  Number of patients experiencing a unfavorable neurological outcome at 12 months, defined as changes in thinking, emotion, will and behavior.
Cognitive deficits | 24 months
  Number of patients experiencing a unfavorable neurological outcome at 24 months, defined as changes in thinking, emotion, will and behavior.
Major adverse cardiac or cerebrovascular events | 10 days after the procedure
  Number of patients experiencing an event including all-cause death, non-fatal cerebrovascular event, non-fatal any myocardial infarction and revascularization at discharge.
Major adverse cardiac or cerebrovascular events | 3 months
  Number of patients experiencing an event including all-cause death, non-fatal cerebrovascular event, non-fatal any myocardial infarction and revascularization at 3 months.
Major adverse cardiac or cerebrovascular events | 6 months
  Number of patients experiencing an event including all-cause death, non-fatal cerebrovascular event, non-fatal any myocardial infarction and revascularization at 6 months.
Major adverse cardiac or cerebrovascular events | 12 months
  Number of patients experiencing an event including all-cause death, non-fatal cerebrovascular event, non-fatal any myocardial infarction and revascularization at 12 months.
Major adverse cardiac or cerebrovascular events | 24 months
  Number of patients experiencing an event including all-cause death, non-fatal cerebrovascular event, non-fatal any myocardial infarction and revascularization at 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Fa Lin, MD, Principal Investigator — Beijing Tiantan Hospital; Yuanli Zhao, MD, Study Chair — Beijing Tiantan Hospital; Jizong Zhao, MD, Study Chair — Beijing Tiantan Hospital; Runting Li, MD, Principal Investigator — Beijing Tiantan Hospital; Xiaolin Chen, MD, Study Director — Beijing Tiantan Hospital; Yu Chen, MD, Principal Investigator — Beijing Tiantan Hospital; Junlin Lu, MD, Principal Investigator — Beijing Tiantan Hospital; Zhipeng Li, MD, Principal Investigator — Beijing Tiantan Hospital; Heze Han, MD, Principal Investigator — Beijing Tiantan Hospital; Debin Yan, MD, Principal Investigator — Beijing Tiantan Hospital; Shuo Wang, MD, Study Chair — Beijing Tiantan Hospital
Locations (2):
- China (2):
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - The First People's Hospital of Neijiang, Neijiang, Sichuan

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) of this study are available from the principal investigator upon reasonable request.
Supporting Information: Study Protocol
Time Frame: 6 months after the study ended
Access Criteria: The IPD of this study are available from the principal investigator upon reasonable request.

REFERENCES:
- [Derived] Tang X, Wang X, Zhu B, Zhou L, Chen X. The prognostic significance of uric acid to albumin ratio in patients with aneurysmal subarachnoid hemorrhage following surgical clipping or endovascular interventions: insights from a large cohort study. Front Neurol. 2026 Jan 12;16:1648805. doi: 10.3389/fneur.2025.1648805. eCollection 2025. PMID 41602990
- [Derived] Yu T, Lau TY, Liu Y, Li R, Lin F, Song Z, Zhu Q, Chen Y, Li T, Jing J, Chen X. Low-Field Portable MRI Detects Developmental Pattern of Ultraearly Cerebral Infarction in aSAH. Stroke. 2025 Dec 11. doi: 10.1161/STROKEAHA.125.052474. Online ahead of print. PMID 41376582
- [Derived] Tang X, Zhu B, Liu M, Lin F, Li R, Song W, Xue J, Zhou L, Chen X. Increased triglyceride-glucose index is associated with adverse functional outcome for patients with aneurysmal subarachnoid hemorrhage after surgical clipping and endovascular coiling: insights from a large cohort study. Front Neurol. 2025 Sep 10;16:1622819. doi: 10.3389/fneur.2025.1622819. eCollection 2025. PMID 41001201
- [Derived] Yang Y, Zhu B, Lin F, Li R, Chen X. Association between geriatric nutritional risk index and clinical outcome of elderly aneurysmal subarachnoid hemorrhage patients: insights from a large cohort study. Neurosurg Rev. 2025 Feb 4;48(1):169. doi: 10.1007/s10143-025-03209-6. PMID 39903290
- [Derived] Li R, Lin F, Chen Y, Lu J, Yang J, Han H, Yuan K, Wang K, Yan D, Li R, He S, Li Z, Zhang H, Chen X, Ma L, Zhao Y, Hao Q, Ye X, Wang H, Li H, Zhang L, Shi G, Zhou J, Li Y, Wang S, Chen X, Zhao Y. The effect of sex differences on complications and 90-day outcomes after aneurysmal subarachnoid hemorrhage: a propensity score-matched analysis. Neurosurg Rev. 2022 Oct;45(5):3339-3347. doi: 10.1007/s10143-022-01836-x. Epub 2022 Jul 23. PMID 35870093
- [Derived] Li R, Lin F, Chen Y, Lu J, Han H, Ma L, Zhao Y, Yan D, Li R, Yang J, He S, Li Z, Zhang H, Yuan K, Wang K, Hao Q, Ye X, Wang H, Li H, Zhang L, Shi G, Zhou J, Zhao Y, Zhang Y, Li Y, Wang S, Chen X, Zhao Y. A 90-Day Prognostic Model Based on the Early Brain Injury Indicators after Aneurysmal Subarachnoid Hemorrhage: the TAPS Score. Transl Stroke Res. 2023 Apr;14(2):200-210. doi: 10.1007/s12975-022-01033-4. Epub 2022 May 14. PMID 35567655
- [Derived] Li R, Lin F, Chen Y, Lu J, Han H, Ma L, Zhao Y, Yan D, Li R, Yang J, He S, Li Z, Zhang H, Yuan K, Wang K, Hao Q, Ye X, Wang H, Li H, Zhang L, Shi G, Zhou J, Zhao Y, Zhang Y, Li Y, Wang S, Chen X, Zhao Y. Elevated blood hemoglobin on admission as an independent predictor of unfavorable outcomes in patients with aneurysmal subarachnoid hemorrhage. Neurosurg Rev. 2022 Aug;45(4):2689-2699. doi: 10.1007/s10143-022-01780-w. Epub 2022 Apr 2. PMID 35366711
- [Derived] Yang J, Lu J, Li R, Lin F, Chen Y, Han H, Yan D, Li R, Li Z, Zhang H, Yuan K, Li H, Zhang L, Shi G, Zhou J, Wang S, Zhao Y, Chen X. Application of Intracranial Pressure-Directed Therapy on Delayed Cerebral Ischemia After Aneurysmal Subarachnoid Hemorrhage. Front Aging Neurosci. 2022 Mar 14;14:831994. doi: 10.3389/fnagi.2022.831994. eCollection 2022. PMID 35360218
- [Derived] Lin F, Chen Y, He Q, Zeng C, Zhang C, Chen X, Zhao Y, Wang S, Zhao J. Prognostic Value of Elevated Cardiac Troponin I After Aneurysmal Subarachnoid Hemorrhage. Front Neurol. 2021 May 31;12:677961. doi: 10.3389/fneur.2021.677961. eCollection 2021. PMID 34135855